CLINICAL TRIAL: NCT05677659
Title: A Phase 2 Safety, Tolerability, and Proof-of-Concept Study of VGL101 in Patients With Adult-Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia (ALSP) (The Ignite Study)
Brief Title: A Study of VGL101 in Patients With Adult-Onset Leukoencephalopathy With Axonal Spheroids and Pigmented Glia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No beneficial effects on biomarker or clinical efficacy endpoints
Sponsor: Vigil Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGL101-01.201
Record Dates: First submitted 2022-11-30; First posted 2023-01-10 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: ALSP
Keywords: ALSP; CSF1R; leukoencephalopathy; Hereditary Diffuse Leukoencephalopathy with Spheroids; HDLS; CSF1R-related Leukoencephalopathy; Adult-Onset Leukoencephalopathy with Axonal Spheroids and Pigmented Glia; CSF1R gene mutation; IGNITE
MeSH Terms: conditions — Leukoencephalopathies; Hereditary Diffuse Leukoencephalopathy with Spheroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VGL101 (Experimental): Solution administered via Intravenous Infusion (IV)
  Interventions: Drug: VGL101

INTERVENTIONS:
Drug: VGL101 — Solution administered via Intravenous Infusion (IV)

SUMMARY:
This is a multicenter, open-label study to assess the safety and tolerability of iluzanebart (also referred to as VGL101) in subjects with documentation of a gene mutation in the CSF1R gene for the treatment of adult-onset leukoencephalopathy with axonal spheroids and pigmented glia (ALSP) and to evaluate the effects of iluzanebart on imaging and biomarkers of disease progression in subjects with ALSP. Participants will receive infusions of iluzanebart approximately every 4 weeks for 1 year. The study includes a 52-week, open-label Core Study, followed by a Long-Term Extension (LTE), which provides subjects who complete the original 52-week study (Core Study) with the option to continue treatment for up to an additional 2 years.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who have documentation of a gene mutation in the CSF1R gene
* Participants fulfill both (Parts A and B) of the following criteria:

  1. The participant has more than 2 findings of clinical signs or symptoms in the following categories:

     1. Cognitive impairment or psychiatric problem
     2. Pyramidal signs on neurological examination
     3. Extrapyramidal signs, such as rigidity.
     4. Epilepsy
  2. MRI findings consistent with ALSP, specifically, bilateral cerebral white matter lesions with or without thinning of the corpus callosum, on the Screening MRI.
* The participant must have a study partner (i.e., caregiver, family member, friend, etc.) who, in the investigator's judgment, has frequent and sufficient contact with the subject so as to be able to provide accurate information about the participant's health and cognitive and functional abilities. The study partner must be willing to sign a study partner ICF.

Key Exclusion Criteria:

* The participant has any neurological disease that poses a risk to the participant or can produce cognitive, motor, or behavioral impairment similar to ALSP, including, but not limited to, brain tumor, hydrocephalus, Alzheimer's disease, frontotemporal dementia (FTD), ALS, stroke, Huntington disease, multiple sclerosis, Parkinson's disease, and Down syndrome.
* Participant with any condition or situation that, in the opinion of the investigator or sponsor medical personnel, may place the subject at significant risk, confound the study results, or interfere significantly with the participant's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Core Study Adverse Events | Through Week 52
  To evaluate the safety and tolerability of iluzanebart for the treatment of adult-onset leukoencephalopathy with axonal spheroids and pigmented glia (ALSP) by adverse events in the Core Study
Long-Term Extension Adverse Events | Week 52 through Week 148
  To evaluate the safety and tolerability of iluzanebart for the treatment of ALSP by adverse events in the Long-Term Extension

SECONDARY OUTCOMES:
To evaluate the effects of iluzanebart on brain volume loss on MRI in subjects with ALSP in the Core Study | Baseline and Week 52
  Percentage of subjects with minimal radiological progression from Baseline to Week 52
To assess the correlation between brain volume loss on MRI and clinical measures of disease progression in subjects with ALSP in the Core Study | Baseline and Week 52
  * Correlation between brain volume loss and Montreal Cognitive Assessment (MoCA) changes from Baseline to Week 52
  * Correlation between brain volume loss and Cortical basal ganglia functional scale (CBFS) changes from Baseline to Week 52
To evaluate the effects of iluzanebart on clinical measures of disease progression in subjects with ALSP in the Core Study | Baseline and Week 52
  * Percentage of subjects with minimal progression in the MoCA scale, from Baseline to Week 52
  * Percentage of subjects with minimal progression in CBFS from Baseline to Week 52
  * Percentage of subjects who did not worsen in the Clinical Global Impression - Change (CGI-C) scale at Week 52
To evaluate the effects of iluzanebart on fluid biomarkers of neurodegeneration in subjects with ALSP in the Core Study | Baseline and Week 52
  Change from Baseline to Week 52 in neurofilament light chain (NfL) in and blood
To evaluate the pharmacokinetics of iluzanebart in subjects with ALSP in the Core Study | Through Week 52
  Serum and cerebrospinal fluid (CSF) concentrations of iluzanebart
To evaluate the effects of iluzanebart on brain volume loss on MRI in subjects with ALSP in the Long-Term Extension | Baseline and Weeks 76, 100, 124, and 148
  Change from Baseline to Weeks 76, 100, 124, and 148 in brain volume loss
To assess the correlation between brain volume loss on MRI and clinical measures of disease progression in subjects with ALSP in the Long-Term Extension | Baseline and Weeks 76, 100, 124, and 148
  * Correlation between brain volume loss and MoCA changes from Baseline to Weeks 76, 100, 124, and 148
  * Correlation between brain volume loss and CBFS changes from Baseline to Weeks 76, 100, 124, and 148
To evaluate the effects of iluzanebart on clinical measures of disease progression in subjects with ALSP in the Long-Term Extension | Baseline and Weeks 64, 76, 88, 100, 112, 124, 136, and 148
  * Change from baseline to Weeks 64, 76, 88, 100, 112, 124, 136, and 148 in the MoCA and CBFS
  * Mean CGI-C score at Weeks 64, 76, 88, 100, 112, 124, 136, and 148
To evaluate the effects of iluzanebart on fluid biomarkers of neurodegeneration in subjects with ALSP in the Long-Term Extension | Baseline and Weeks 76, 100, 124, and 148
  Change from Baseline to Weeks 76, 100, 124, and 148 in NfL in blood
To evaluate the pharmacokinetics of iluzanebart in subjects with ALSP in the Long-Term Extension | Week 52 through Week 148
  Serum and CSF concentrations of iluzanebart

CONTACTS AND LOCATIONS:
Locations (10):
- United States (5):
  - Investigative Site 3, San Francisco, California
  - Investigative Site 2, Englewood, Colorado
  - Investigative Site 1, Jacksonville, Florida
  - Investigative Site 5, Boston, Massachusetts
  - Investigative Site 6, Philadelphia, Pennsylvania
- Investigative Site 10, Paris, France
- Germany (2):
  - Investigative Site 7, Leipzig
  - Investigative Site 9, Tübingen
- Investigative Site 8, Amsterdam, Netherlands
- Investigative Site 4, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No